CLINICAL TRIAL: NCT06444243
Title: A Multi-centre, Double-blinded, Placebo-controlled, Randomised, Phase II Clinical Trial for Psilocybin-assisted Therapy for Alcohol Use Disorder
Brief Title: Psilocybin-assisted Therapy for Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Woke Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: X23-0055
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Depression; Anxiety
Keywords: Psilocybin-assisted therapy; Randomised-Controlled Trial; Psilocybin; Psychedelic-Assisted Therapy; Alcohol Use Disorder Therapy
MeSH Terms: conditions — Alcoholism; Depression; Anxiety Disorders | interventions — Psilocybin; Niacin

STUDY DESIGN:
Intervention Model Description: Multi-centre, Double-blinded, Randomised, Phase II Clinical Trial for Psilocybin-assisted Therapy for Alcohol Use Disorder
Who Masked: Participant, Care Provider
Masking Description: Double blinded with an additional optional dosing session for open label dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Psilocybin + Therapy (Experimental): * 12 weekly sessions of psychotherapy for AUD
  * 2 dosing sessions - psilocybin 25mg
  * Additional open-label dosing session for participants in control arm post-follow up
  * 2 integration sessions following each dosing session (additional dosing session for open label dosing)
  * 3 post-treatment follow-up sessions
  * Total of 13 clinic sessions
  Interventions: Drug: Psilocybin
- Niacin + Therapy (Placebo Comparator): * 12 weekly sessions of psychotherapy for AUD
  * 2 dosing sessions - niacin 250mg
  * 2 integration sessions following each dosing session
  * 3 post-treatment follow-up sessions
  * Total of 13 clinic sessions
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a naturally occurring psychedelic prodrug compound produced by more than 200 species of fungi.
  Arms: Psilocybin + Therapy
Drug: Niacin — A nutrient in the vitamin B complex that the body needs in small amounts to function and stay healthy. Niacin helps some enzymes work properly and helps skin, nerves, and the digestive tract stay healthy. Niacin is found in many plant and animal products.
  Niacin will be used at a concentration of 250mg as an active control.
  Arms: Niacin + Therapy

SUMMARY:
To explore the effectiveness of psilocybin-assisted therapy on reducing alcohol consumption in a double-blind, randomised, phase II clinical trial.

DETAILED DESCRIPTION:
New strategies for treating Alcohol Use Disorder (AUD) are urgently needed. Recent evidence has shown promising results for psychedelic-assisted therapies, particularly psilocybin, which has demonstrated efficacy in reducing alcohol consumption and improving psychological well-being. This study aims to evaluate the clinical efficacy and tolerability of psilocybin-assisted therapy compared to a control (niacin) in reducing heavy drinking days (HDD) per week among individuals with AUD.

Primary Objective

To conduct a double-blind, randomised controlled trial with 90 participants diagnosed with Alcohol Use Disorder (AUD). The primary aim is to compare the efficacy of psilocybin-assisted therapy (two sessions of psilocybin, 25 mg per dosing session) versus control (niacin 250mg) and therapy in reducing alcohol consumption, specifically measuring the number of heavy drinking days (HDD) per week.

Secondary Objectives

To compare the efficacy of psilocybin-assisted therapy versus control in improving the characteristics of AUD and addressing common comorbidities associated with AUD, including depression and anxiety.

Study Design

The trial will employ a double-blind, randomised, controlled design. A sample of 90 individuals with AUD will undergo 14 weeks of treatment, which includes 12 therapy sessions and 2 dosing sessions with either psilocybin (25 mg) or control (niacin 250mg). Participants will be assessed for changes in alcohol consumption patterns and improvements in symptoms of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe AUD according to the DSM-5 criteria
2. A desire to reduce or stop drinking
3. Consumed at least 21 standard drinks per week or ≥2 HDD (≥5 standard drinks/day for men; ≥4 for women) in the past week prior to screening
4. Aged ≥18 years old
5. Adequate cognition and English language skills to give valid consent and complete research interviews and assessments (MoCA ≥26)
6. Received prior treatment for AUD (not including study interventions)
7. Stable housing within reasonable distance to a clinical site for the duration of the study
8. Able to identify a significant other (such as a family/friend/partner) who could accompany them from clinic/provide transport and/or be contacted by the study team if required
9. Willing to give written informed consent

Exclusion Criteria:

* a. History of or currently meeting DSM-5 criteria for:

  * Any psychotic disorder
  * Bipolar disorder type 1 or 2
  * Major depression with psychotic features
  * Any personality disorders
  * Post-traumatic stress disorder
  * Hallucinogen persisting perception disorder b. A family history of:
  * Schizophrenia or schizoaffective disorder (first- or second-degree relatives), or
  * Bipolar disorder type 1 (first degree relatives) c. Suicide risk according to clinician judgement (e.g. previous suicide attempt or self-harm in the past 6 months) and responses to Columbia Suicide Severity Rating Scale (C-SSRS) and SCID-5-RV.

    d. Abnormal and/or serious clinical finding or medical condition that may preclude participation e. Concurrent use of psychotropic medication e.g., antidepressants, antipsychotics, psychostimulants, treatments for addictions, other dopaminergic or serotonergic agents (e.g. St John's Wort/tryptophan), lithium, anticonvulsants).
  * Use of antidepressants and alcohol pharmacotherapy use considered if assessed by investigator and titrated down with 5 half-lives + 1-week washout f. Use of any medications likely to interact with study medication during the trial (subject to investigator's discretion).
  * Low dose opiates permitted for pain management, however, not the night before or after dosing sessions g. Significant alcohol withdrawal (current CIWA-Ar score ≥10, including history of delirium tremens or alcohol withdrawal seizures).

    h. Any current substance use disorder (SUD) other than tobacco (e.g. opiates, benzodiazepines, cannabis, psychostimulants, hallucinogens) as per clinician judgement and/or defined by DSM-5 criteria (measured by SCID-RV).

    i. Substantial lifetime use (>25 total) or recent use (past 12 months) of ketamine or classic hallucinogens, such as psilocybin-containing mushrooms or LSD j. Any alcohol pharmacotherapy (e.g. naltrexone, acamprosate) within the past month.

    k. Participation in other clinical trials in the previous two months l. Pregnant or lactating (contraception must be used and a sensitive pregnancy test will be performed at baseline and prior to dosing) m. Allergy or hypersensitivity to psilocybin n. Any condition or factor deemed by the study clinician to place the individual at higher risk of an adverse emotional reaction, severe active stressors such as significant legal problems, marital distress or lack of social support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Heavy Drinking Days (HDD) | 52 Weeks
  Frequency of HDD as measured by the Timeline Follow Back (TLFB) and validated by Phosphatidylethanol (PEth). HDD are defined as ≥4 drinks/day for women and ≥5 drinks/day for men.

SECONDARY OUTCOMES:
Mean alcohol consumption per drinking day | 52 Weeks
  The mean alcohol consumption per drinking day will be gathered reported as the number of standard drinks consumed each day.
Absence of any HDD | 52 Weeks
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
WHO drinking risk level | 52 Weeks
  The WHO categorizes alcohol consumption into different risk levels based on average daily intake and associated health risks: Abstainer: Rarely or never drinks alcohol. Low-risk drinking: (Men: Up to 2 standard drinks per day, Women: Up to 1 standard drink per day). Moderate-risk drinking: (Men: 3-4 standard drinks per day, Women: 2-3 standard drinks per day). High-risk drinking: (Men: More than 4 standard drinks per day, Women: More than 3 standard drinks per day). Heavy episodic (binge) drinking: 60 grams (5-6 drinks) or more on a single occasion.
Dependence Severity | 52 Weeks
  Alcohol Dependence Scale (ADS) is a measure of the severity of the participant's dependence on alcohol. The measure contains 29 items regarding symptoms and occurrences associated with dependence on alcohol. A total score for the measure is yielded by adding across items. Higher scores indicate more severe dependence.
Alcohol Craving | 52 Weeks
  Alcohol craving will be investigated using the Penn Alcohol Craving Scale (PACS). The PACs is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week.
PEth Levels | 52 Weeks
  PEth measures the level of phosphatidylethanol, a direct alcohol biomarker which is found in human blood following alcohol consumption. Phosphatidylethanols are abnormal phospholipids formed in the presence of ethanol
Changes in Anxiety | 52 Weeks
  Measured by cumulative scores on the DASS-21 Anxiety Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more anxiety.
Changes in Depression | 52 Weeks
  Measured by cumulative scores on the DASS-21 Depression Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates greater depression.
Changes in Suicidal Ideation | 52 Weeks
  Changes in suicidal ideation & behaviours across the treatment period. This will be measured on the C-SRSS (Columbia Suicide Severity Rating Scale). At baseline this will be measured by the baseline version. At each visit following this, this will be recorded on the since last visit version. Higher scores indicate more severe suicidality.
Changes in Quality of Life | 52 Weeks
  To assess whether treatment can change quality of life as measured by the short form Health Survey (SF-36). This survey has 36 items that measure 8 domains of health, including: physical functioning, physical role limitations, bodily pain, general health perceptions, energy/vitality, social functioning, emotional role limitations and mental health. The scores are transformed to range from 0 (worst possible health) to 100 (best possible health).
Markers of Liver Injury | 52 Weeks
  An assortment of liver enzymes will be monitored throughout the trial to investigate any changes that occur in liver function.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haber, PhD, Principal Investigator — University of Sydney; Kirsten C Morley, PhD, Principal Investigator — University of Sydney

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) might not be shared due to privacy concerns, potential misuse of data, intellectual property rights, and ethical considerations. Additionally, legal restrictions and the need to protect sensitive information can also limit the sharing of IPD.